CLINICAL TRIAL: NCT02685072
Title: Progesterone Augmentation of Nicotine Replacement Therapy Study
Acronym: PANS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1504015618; R21CA198187 (NIH)
Record Dates: First submitted 2015-12-17; First posted 2016-02-18 (Estimated); Results first posted 2019-07-23 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Smoking Cessation
Keywords: Smoking Cessation; Nicotine Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Progesterone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TNP + Progesterone (Experimental): Transdermal Nicotine Patch + Progesterone (200 mgs BID)
  Interventions: Drug: Progesterone (200 mgs BID)
- TNP + Placebo (Placebo Comparator): Transdermal Nicotine Patch + Placebo (for Progesterone)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Progesterone (200 mgs BID) — Transdermal Nicotine Patch (TNP) + Progesterone
  Other Names: Prometrium
  Arms: TNP + Progesterone
Drug: Placebo — TNP + Placebo
  Arms: TNP + Placebo

SUMMARY:
This will be a double-blind, placebo-controlled, pilot, randomized clinical trial. A total of 50 women who smoke and have regular menstrual cycles will be randomized to either progesterone (200 mgs BID) + Transdermal Nicotine Patch (TNP) or placebo + TNP for 8 weeks. TNP will be tapered after 4-6 weeks. Progesterone or matching placebo will be discontinued at the end of Week 8. All participants will also be provided behavioral treatment for smoking cessation. Participants will be inducted onto progesterone (or placebo) + TNP over a one-week period (Week 1) during the mid luteal phase, within a week before menses and the target quit date will be set for the 5 (+/-2) days after onset of menses. Participants will have post-trial follow-up visits at 1 and 3 months.The main study outcomes will be self- report of smoking abstinence, biochemically verified smoking abstinence, measures of cigarette craving and nicotine withdrawal, and measures of response inhibition.

DETAILED DESCRIPTION:
This study seeks to determine if modifying the hormonal milieu of the menstrual cycle, through administration of exogenous progesterone, will improve the effectiveness of treatments for smoking cessation in women. Progesterone, a gonadal hormone, is used clinically for treatment of endometrial hyperplasia, amenorrhea, dysfunctional uterine bleeding, and for assisted reproduction in women. Progesterone also shows promise for the treatment of multiple central nervous system disorders including cocaine addiction, seizure disorder, and traumatic brain injury. As the next step, the investigators seek to determine if progesterone augments standard smoking cessation treatments (e.g., NRT) in regularly cycling women. The investigators hypothesize that co-treatment with progesterone, compared to placebo, will enhance the effectiveness NRT for smoking cessation. To test this hypothesis, the investigators propose an 8-week, double-blind, placebo-controlled clinical trial, which will randomize 50 smokers using a 1:1 assignment ratio to 400 mg/day progesterone or placebo. Consistent with the Clinical Practice Guidelines, all participants will also receive transdermal nicotine patch (TNP) plus brief counseling for smoking cessation during the study participation.

Specific Aim #1: To determine if progesterone +TNP is superior to placebo +TNP for prolonged and 7-day point prevalence of smoking abstinence rates at the end of 8 weeks of treatment and at 1 and 3 month follow-up time points. The investigators will also evaluate the safety and tolerability of progesterone treatment, compared to placebo. Our co-primary outcome measures will be 7-day point prevalence of smoking abstinence and breath CO at the end of treatment and 1- and 3-months after the end of the trial. Specific Aim #2: To determine if progesterone + TNP treatment, compared to placebo + TNP, improves response inhibitory function, as assessed by the Stroop, The Go/No Go task, and the Digit Symbol Task. Specific Aim # 3: To determine if progesterone + TNP treatment, compared to placebo + TNP, leads to a greater reduction in cigarette craving and nicotine withdrawal symptoms, as assessed by the Questionnaire on Smoking Urges-Brief (QSU-B) and the Minnesota Nicotine Withdrawal Scale (MNWS), respectively. Specific Aim #4: To evaluate with affective changes, as shown on the Positive and Negative Affect Schedule, mediates the effects of progesterone on smoking abstinence.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 - 45
* Smoking at least 5 cigarettes/ day for at least one year
* Regular menstrual cycles every 24-36 days for the previous 6 months
* Motivated to quit smoking (i.e., a rating of at least "7 "on a 10-point scale where 1 is not at all motivated and 10 is extremely motivated)
* In good health
* Using an acceptable, non-hormonal birth control

Exclusion Criteria:

A history of major medical or psychological illnesses including:

* liver disease
* heart disease
* diabetes
* malignancy including history of breast cancer
* deep vein thrombosis
* blood coagulation problems including a history or family history of thrombophilia
* liver failure
* cervical intra-epithelial lesions III or greater that are untreated
* other medical conditions that the physician investigators deems will make study participation unsafe for the subject
* current or past history bipolar disorder or schizophrenia
* current diagnosis of major depression
* panic disorder or post-traumatic stress disorder
* active drug (non-nicotine) and/or alcohol dependence
* currently undergoing treatment with another pharmacological agent for smoking cessation
* regular use of sedating medications including sleeping aids, antihistamines, and others use of nicotine from cigars, pipes, chewing tobacco
* pregnant
* breast- feeding or intending to become pregnant within 6 months
* allergy to nicotine patch or progesterone
* allergy to peanuts or other nuts.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2016-04-07 (Actual); Primary Completion 2017-12-18 (Actual); Study Completion 2018-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Yonkers, MD, Principal Investigator — Yale University
Locations (1):
- Yale School of Medicine, Department of Psychiatry, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
we will only make aggregate de-identified data available

RESULTS

PARTICIPANT FLOW:
Groups:
- TNP + Progesterone: Transdermal Nicotine Patch + Progesterone (200 mgs BID)
  Progesterone (200 mgs BID): TNP + Progesterone
Period: Treatment Period
Arm/Group | TNP + Progesterone | TNP + Placebo
Started | 33 | 31
Completed Week 2 Visit | 23 | 26
Completed Week 3 Visit | 20 | 23
Completed Week 4 Visit | 19 | 23
Completed Week 5 Visit | 19 | 22
Completed Week 6 Visit | 18 | 19
Completed Week 7 Visit | 17 | 18
Completed Week 8 Visit (End of study treatment period) | 20 | 22 (Week 8 data were collected at the 1-month follow-up for 1 participant)
Completed | 20 | 22
Not Completed | 13 | 9
Not completed — Lost to Follow-up | 12 | 6
Not completed — Withdrawal by Subject | 1 | 3
Period: 1-Month Follow-Up
Arm/Group | TNP + Progesterone | TNP + Placebo
Started | 20 | 22
Completed | 19 | 22
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: 3-Month Follow-Up
Arm/Group | TNP + Progesterone | TNP + Placebo
Started | 19 | 22
Completed | 19 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TNP + Progesterone | TNP + Placebo | Total
Number analyzed (Participants) | 33 | 31 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.3 (7.6) | 33.0 (8.0) | 32.6 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 31 | 64
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 4 | 12
  Not Hispanic or Latino | 24 | 27 | 51
  Unknown or Not Reported | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 14 | 21 | 35
  White | 12 | 9 | 21
  MIxed Race | 6 | 1 | 7
  unknown | 1 | 0 | 1
Cigarettes per day [Mean (Standard Deviation); unit: cigarettes per day] | 11.4 (7.0) | 13.2 (7.3) | 12.3 (7.2)
Motivation to quit smoking [Mean (Standard Deviation); unit: units on a scale] — Participants were asked on a scale from 1 (not motivated at all) to 10 (extremely motivated), how motivated are you to quit smoking?
  units on a scale | 9.0 (1.1) | 8.9 (1.3) | 8.9 (1.2)
Lives with smoker [Count of Participants; unit: Participants]
  Lives with smoker | 19 | 19 | 38
  Does not live with smoker | 14 | 12 | 26

OUTCOME MEASURES:

1. Primary Outcome: 7-day Point Prevalence of Smoking Abstinence
Description: The 7-day point prevalence is defined by self-reported smoking abstinence for the last 7 days.
Time Frame: end of 8 weeks of treatment
Population: Participants (n=13 in TPN + Progesterone; n=9 in TPN + Placebo) missing outcome data were coded as not abstinent.
Measure: Count of Participants; unit: Participants
Arm/Group | TNP + Progesterone | TNP + Placebo
Number analyzed (Participants) | 33 | 31
Participants
  abstinent | 8 | 11
  not abstinent | 25 | 20
Statistical Analysis 1: Comparison: TNP + Progesterone vs TNP + Placebo; Test type: Superiority; p = 0.3253, Chi-squared; degrees of freedom =1; Odds Ratio (OR) = 0.5818, 95% CI 2-sided [0.1968 to 1.7202] — Odds ratio represents odds of smoking abstinence in TPN + progesterone group versus TPN + placebo group

2. Secondary Outcome: Carbon Monoxide <10 Ppm
Description: Smoking abstinence measured by breath CO
Time Frame: end of 8 weeks of treatment
Population: Participants (n=13 in TPN + Progesterone; n=10 in TPN + Placebo) missing breath CO were coded as ≥ 10 ppm (positive for smoking).
Measure: Count of Participants; unit: Participants
Arm/Group | TNP + Progesterone | TNP + Placebo
Number analyzed (Participants) | 33 | 31
Participants
  CO <10 ppm | 9 | 8
  CO ≥ 10 ppm | 24 | 23
Statistical Analysis 1: Comparison: TNP + Progesterone vs TNP + Placebo; Test type: Superiority; p = 0.8944, Chi-squared; degrees of freedom = 1; Odds Ratio (OR) = 1.0781, 95% CI 2-sided [0.3550 to 3.2744] — Odds ratio represents odds of CO < 10 (negative for smoking) in TPN + progesterone versus TPN + placebo groups

3. Secondary Outcome: Carbon Monoxide <10 Ppm
Description: Smoking abstinence measured by breath CO
Time Frame: 1 month follow up
Population: Participants (n=14 in TPN + progesterone; n=9 in TPN + placebo) missing breath CO data were coded as > 10 ppm (positive for smoking).
Measure: Count of Participants; unit: Participants
Arm/Group | TNP + Progesterone | TNP + Placebo
Number analyzed (Participants) | 33 | 31
Participants
  CO <10 ppm | 6 | 7
  CO ≥ 10 ppm | 27 | 24
Statistical Analysis 1: Comparison: TNP + Progesterone vs TNP + Placebo; Test type: Superiority; p = 0.6620, Chi-squared; degrees of freedom = 1; Odds Ratio (OR) = 0.7619, 95% CI 2-sided [0.2247 to 2.5838] — Odds ratio represents odds of CO < 10 ppm (negative for smoking) in TPN + progesterone versus TPN + placebo

4. Secondary Outcome: Carbon Monoxide <10 Ppm
Description: Smoking abstinence measured by breath CO
Time Frame: 3 month follow up
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | TNP + Progesterone | TNP + Placebo
Number analyzed (Participants) | 33 | 31
Participants
  CO <10 ppm | 10 | 10
  CO ≥ 10 ppm | 23 | 21
Statistical Analysis 1: Comparison: TNP + Progesterone vs TNP + Placebo; Test type: Superiority; p = 0.8661, Chi-squared; degrees of freedom = 1; Odds Ratio (OR) = 0.9130, 95% CI 2-sided [0.3171 to 2.6287] — Odds ratio represents odds of CO < 10 ppm (negative for smoking) in TPN + progesterone versus TPN + placebo

5. Secondary Outcome: Change in Stroop Measure of Inhibitory Function
Description: The Stroop test assesses cognitive processing. The Level 3 Stroop Throughput score incorporates both accuracy and speed. In Level 3 of the Stroop test, a series of words representing colors are shown in a font color that is incongruent with the word (e.g. RED would be shown in blue font). Users are asked to press a response key associated with the color of the font, not the written word. Quicker and more accurate responses lead to higher scores. The lowest possible score is 0 (no correct responses). There is no defined maximum score, as the score depends upon both response time and number of correct responses. A Level 3 Stroop Throughput change score was calculated by subtracting baseline score from week 2 score. Higher positive scores represent greater improvement in scores at week 2 relative to baseline, and lower negative scores represent greater decline in scores from baseline to week 2.
Time Frame: baseline and week 2
Population: Includes people who completed Stroop Test at both baseline and Week 2 visits.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TNP + Progesterone | TNP + Placebo
Number analyzed (Participants) | 24 | 26
units on a scale | 4.1 (24.7) | -5.0 (28.7)
Statistical Analysis 1: Comparison: TNP + Progesterone vs TNP + Placebo; Test type: Superiority; p = 0.31, t-test, 2 sided; Mean Difference (Final Values) = -9.1, 95% CI 2-sided [-27.1 to 9.0], Standard Deviation 31.7 — (Placebo + TPN) - (Progesterone + TPN)

6. Secondary Outcome: Change in Go/No Go Task Measure of Inhibitory Function
Description: Week 2 minus baseline. This task assesses the ability to withhold responses to an infrequently occurring target (No-Go trials). A total of 225 single digits (25 x 9 digits) are presented on a computer monitor for 250 ms each, immediately followed by a mask for 900 ms. Subjects must press a spacebar in response to every digit except the "3".
  Go/No Go score is calculated as separation between the means of the signal and the noise distributions and is reported in standard deviation units, representing an overall indicator of performance since it accounts for correct responses and incorrect responses. Higher scores represent a better outcome. For the change score, higher positive scores represent greater improvement in scores between baseline and week 2, and lower negative scores represent greater decline in scores between baseline and week 2.
Time Frame: baseline and week 2
Population: Includes participants who completed the Go/No Go task at both baseline and week 2 visits.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TNP + Progesterone | TNP + Placebo
Number analyzed (Participants) | 24 | 26
units on a scale | 0.36 (2.33) | 0.50 (1.45)
Statistical Analysis 1: Comparison: TNP + Progesterone vs TNP + Placebo; Test type: Superiority; p = 0.7910, t-test, 2 sided; Mean Difference (Final Values) = 0.1480, 95% CI 2-sided [-0.9747 to 1.2707] — (placebo + TPN) - (progesterone + TPN)

7. Secondary Outcome: Change in Digit Symbol Task Measure of Inhibitory Function
Description: The Code Substitution Test (a computerized adaptation/variant of the Digit Symbol Substitution Test) is a test of psychomotor performance. The Code Substitution-Learning Throughput Score incorporates both accuracy and speed. During the learning phase of this test, users are continuously shown a row of 9 digits that are paired with a symbol (the pairings are constant). Users are presented with a series of individual pairings and are asked to press a response key to indicate if the pairing is correct or not. Quicker and more accurate responses lead to higher scores. The lowest possible score is 0 (no correct responses). There is no defined maximum score, as the score depends upon both response time and number of correct responses. A change score was calculated by subtracting baseline score from week 2 score. Higher positive scores represent greater improvement in scores at week 2 relative to baseline, and lower negative scores represent greater decline in scores from baseline to week 2.
Time Frame: baseline and week 2
Population: Includes participants who completed the Code Substitution-Learning Test.at both baseline and week 2 visits.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TNP + Progesterone | TNP + Placebo
Number analyzed (Participants) | 24 | 33
units on a scale | -3.95 (11.42) | 5.32 (11.59)
Statistical Analysis 1: Comparison: TNP + Progesterone vs TNP + Placebo; Test type: Superiority; p = 0.0065, t-test, 2 sided; Mean Difference (Final Values) = 9.26, 95% CI 2-sided [2.71 to 15.81]

8. Secondary Outcome: Positive and Negative Affect Schedule (PANAS) Total Score
Description: The PANAS questionnaire consists of 20 items that describe different feelings and emotions. Participants are asked to what extent they feel this way right now on 5-point scale ranging from 1 (very slightly or not at all) to 5 (extremely). Separate Positive Affect Scores and Negative Affect Scores were calculated from 10 items each. Scores can range from 10 t0 50, with higher scores representing higher levels of positive affect and with lower scores representing lower levels of negative affect.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TNP + Progesterone | TNP + Placebo
Number analyzed (Participants) | 33 | 31
score on a scale
  Positive Affect Score | 29.2 (7.0) | 25.6 (7.7)
  Negative Affect Score | 11.9 (2.1) | 11.4 (1.8)

9. Secondary Outcome: Positive and Negative Affect Schedule (PANAS) Total Score
Description: as for outcome 8
Time Frame: Week 2
Population: Note: numbered analyzed does not equal 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TNP + Progesterone | TNP + Placebo
Number analyzed (Participants) | 23 | 26
score on a scale
  Positive Affect Score | 27.0 (7.1) | 24.4 (8.3)
  Negative Affect Score | 11.4 (1.9) | 11.3 (1.7)

10. Secondary Outcome: Positive and Negative Affect Schedule (PANAS) Total Score
Description: as for outcome 8
Time Frame: Week 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TNP + Progesterone | TNP + Placebo
Number analyzed (Participants) | 20 | 23
score on a scale
  Positive Affect Score | 23.8 (8.6) | 27.0 (8.0)
  Negative Affect Score | 11.6 (2.1) | 12.1 (4.3)

11. Secondary Outcome: Positive and Negative Affect Schedule (PANAS) Total Score
Description: as for outcome 8
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TNP + Progesterone | TNP + Placebo
Number analyzed (Participants) | 19 | 23
score on a scale
  Positive Affect Score | 28.0 (7.4) | 26.3 (9.1)
  Negative Affect Score | 10.6 (1.3) | 11.6 (3.3)

12. Secondary Outcome: Positive and Negative Affect Schedule (PANAS) Total Score
Description: as for outcome 8
Time Frame: Week 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TNP + Progesterone | TNP + Placebo
Number analyzed (Participants) | 19 | 22
score on a scale
  Positive Affect Score | 24.3 (8.6) | 27.9 (9.1)
  Negative Affect Score | 10.7 (1.0) | 10.6 (1.2)

13. Secondary Outcome: Positive and Negative Affect Schedule (PANAS) Total Score
Description: as for outcome 8
Time Frame: Week 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TNP + Progesterone | TNP + Placebo
Number analyzed (Participants) | 18 | 19
score on a scale
  Positive Affect Score | 25.9 (10.0) | 25.7 (10.0)
  Negative Affect Score | 10.9 (1.8) | 11.6 (3.3)

14. Secondary Outcome: Positive and Negative Affect Schedule (PANAS) Total Score
Description: as for outcome 8
Time Frame: Week 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TNP + Progesterone | TNP + Placebo
Number analyzed (Participants) | 17 | 18
score on a scale
  Positive Affect Score | 24.7 (9.1) | 24.7 (9.9)
  Negative Affect Score | 11.5 (3.2) | 10.9 (1.6)

15. Secondary Outcome: Positive and Negative Affect Schedule (PANAS) Total Score
Description: as for outcome 8
Time Frame: Week 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TNP + Progesterone | TNP + Placebo
Number analyzed (Participants) | 20 | 21
score on a scale
  Positive Affect Score | 25.2 (10.4) | 26.5 (10.3)
  Negative Affect Score | 11.6 (2.7) | 10.8 (1.5)

16. Secondary Outcome: Positive and Negative Affect Schedule (PANAS) Total Score
Description: as for outcome 8
Time Frame: 1 month follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TNP + Progesterone | TNP + Placebo
Number analyzed (Participants) | 19 | 22
score on a scale
  Positive Affect Score | 26.4 (8.7) | 26.4 (8.7)
  Negative Affect Score | 10.7 (1.1) | 11.0 (1.7)

17. Secondary Outcome: Positive and Negative Affect Schedule (PANAS) Total Score
Description: as for outcome 8
Time Frame: 3 month follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TNP + Progesterone | TNP + Placebo
Number analyzed (Participants) | 19 | 22
score on a scale
  Positive Affect Score | 24.8 (7.8) | 27.7 (9.2)
  Negative Affect Score | 11.3 (1.6) | 11.1 (1.8)

18. Secondary Outcome: Prolonged Abstinence Post Trial
Description: Abstinence from 2 weeks post quit date to the one month follow up
Time Frame: 1-month follow-up after end of treatment
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | TNP + Progesterone | TNP + Placebo
Number analyzed (Participants) | 33 | 31
Participants
  abstinent | 4 | 5
  not abstinent | 29 | 26
Statistical Analysis 1: Comparison: TNP + Progesterone vs TNP + Placebo; Test type: Superiority; p = .6449, Chi-squared; degrees of freedom = 1; Odds Ratio (OR) = 0.7172, 95% CI 2-sided [0.1738 to 2.9594] — Odds ratio represents odds of CO < 10 ppm (negative for smoking) in TPN + progesterone versus TPN + placebo

19. Secondary Outcome: Prolonged Abstinence Follow up
Description: Abstinence from 2 weeks post quit date to 3 month follow up (total of 6-8 weeks during the trial and 3 month follow up)
Time Frame: 3-month follow-up after end of treatment
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | TNP + Progesterone | TNP + Placebo
Number analyzed (Participants) | 33 | 31
Participants
  abstinent | 4 | 5
  not abstienent | 29 | 26
Statistical Analysis 1: Comparison: TNP + Progesterone vs TNP + Placebo; Test type: Superiority; p = 0.6449, Chi-squared; degrees of freedom = 1; Odds Ratio (OR) = 0.7172, 95% CI 2-sided [0.1738 to 2.9594] — Odds ratio represents odds of prolonged abstinence in TPN + progesterone versus TPN + placebo

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | TNP + Progesterone | TNP + Placebo
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/31
Other Adverse Events (participants affected / at risk) | 4/33 | 4/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TNP + Progesterone (N=33) | TNP + Placebo (N=31)
nausea, vomiting, diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
wrist and back injury due to fall (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
ER visit for unknown reason (General disorders) | 1 (1) | 2 (2)
3 Menses in one month (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-30): https://cdn.clinicaltrials.gov/large-docs/72/NCT02685072/Prot_SAP_000.pdf